CLINICAL TRIAL: NCT00144560
Title: An Open-Label, Clinical Pharmacology Study to Investigate Drug-Drug Interaction in Patients With RA
Brief Title: Drug-Drug Interaction Study of MRA in Patient With Rheumatoid Arthritis (RA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Chugai Pharmaceutical, Chugai Pharmaceutical
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRA220JP
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2008-12-15 (Estimated); Status verified 2008-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

INTERVENTIONS:
Drug: MRA(Tocilizumab)

SUMMARY:
This is an open-label, clinical pharmacology study to investigate drug-drug interaction in patients with RA.

ELIGIBILITY:
Inclusion criteria

* Patients who are diagnosed with RA according to the 1987 American College of Rheumatology (ACR) classification criteria
* Patients who contracted RA at least 6 months prior

Exclusion criteria

* Patients with Class IV Steinbrocker functional impairment at enrollment.
* Patients who have been treated for the underlying disease with a biological agent, such as infliximab or etanercept and have been receiving treatment with leflunomide, within 12 weeks before initiation of treatment with the probe drug

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-02; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
20% improvement based on the ACR criteria compared with the baseline value. | throughout study

SECONDARY OUTCOMES:
Time courses taken from baseline values for DAS28, for ACR20%, 50%, and 70% improvement, and for each ACR core set variable. | Week 0,Week 1, Week 2

CONTACTS AND LOCATIONS:
Overall Officials: Takahiro Kakehi, Study Director — Chugai Pharmaceutical